CLINICAL TRIAL: NCT07027059
Title: The Effect of Neural Mobilization Exercises on Pain and Central Sensitization in Individuals With Lateral Epicondylitis: A Randomized Controlled Trial
Brief Title: Neural Mobilization Exercises on Pain and Central Sensitization
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, kevser kacmaz, research asisstant, phd, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Lepicondilitis
Record Dates: First submitted 2025-06-02; First posted 2025-06-18 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Lateral Epicondylitis
Keywords: lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mobilization (Experimental): participants will receive additional median nerve mobilizations
  Interventions: Behavioral: median nerve mobilization; Behavioral: routine exercises for lateral epicondylisits
- control (Active Comparator): participants will receive routine exercises
  Interventions: Behavioral: routine exercises for lateral epicondylisits

INTERVENTIONS:
Behavioral: median nerve mobilization — An exercise to increase median nerve mobility by flexing and extending fingers, wrist, elbow, shoulder, and neck
  Arms: mobilization
Behavioral: routine exercises for lateral epicondylisits — eccentric strengthening exercises

SUMMARY:
This study aims to investigate the effects of neural mobilization exercises on central sensitization and pain characteristics in individuals with lateral epicondylitis. Enrolled participants will be randomly assigned to two groups. One group will receive routine exercises and ESWT treatment, while the other group will receive neural mobilization exercises in addition to routine exercises and ESWT treatment.

DETAILED DESCRIPTION:
This study aims to investigate the effects of neural mobilization exercises on central sensitization and pain characteristics in individuals with lateral epicondylitis. Enrolled participants will be randomly assigned to two groups. One group will receive routine exercises and ESWT treatment, while the other group will receive neural mobilization exercises in addition to routine exercises and ESWT treatment.

Median nerve mobilizations will be implemented as the neural mobilization exercises. All groups will receive two sessions per week and complete the process in four weeks; therefore, they will have received a total of eight sessions by the end of the study. Routine exercises and median nerve mobilizations will be implemented in every session (twice a week), while ESWT will be implemented once a week.

Median nerve mobilizations will be administered in 5 sets, each consisting of 10 repetitions per session.

Before and after the sessions, subjective factors related to pain will be assessed using the Central Sensitization Scale and the Pain Catastrophizing Scale, as well as pressure pain threshold measurements.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of lateral epicondylitis
* 18-65 years old

Exclusion Criteria:

Any other pathology, disease, condition, pain, surgery on the elbow, wrist, fingers, shoulder, or neck in the last year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Central Sensitization | baseline and after the 8 sessions (4th week)
  pressure pain threshold

SECONDARY OUTCOMES:
Central Sensitization | baseline and after the 8 sessions (4th week)
  Central Sensitization scale
Pain Catastrophizing | baseline and after the 8 sessions (4th week)
  Pain Catastrophizing scale

CONTACTS AND LOCATIONS:
Overall Officials: kevser sevik kacmaz, pt, phd, Principal Investigator — Izmir Katip Celebi University
Locations (1):
- Izmir Katip Celebi University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coombes BK, Bisset L, Vicenzino B. Management of Lateral Elbow Tendinopathy: One Size Does Not Fit All. J Orthop Sports Phys Ther. 2015 Nov;45(11):938-49. doi: 10.2519/jospt.2015.5841. Epub 2015 Sep 17. PMID 26381484